CLINICAL TRIAL: NCT06010732
Title: Comparison of the Remineralization Potential of an Optimized Fluoride Dentifrice With a Control Fluoride Dentifrice Using an in Situ Caries Model
Brief Title: In Situ Comparison of the Remineralization Potential of Optimized Fluoride Dentifrice With Control Fluoride Dentifrice
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: HALEON (Industry)
Responsible Party: Principal Investigator, Domenick Zero, Principal Investigator, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 23-I-121
Record Dates: First submitted 2023-08-17; First posted 2023-08-25 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Caries
Keywords: Caries; Remineralization; Fluoride; Dentifrice
MeSH Terms: interventions — Sodium Fluoride; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Test-Positive-Placebo (Other): Crossover design - Cleaning, 2-3 day non-Fluoride (F) dentifrice, Period 1 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 2 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 3 product for 2 weeks. Product sequence: 1100 ppm F as sodium fluoride Test Product,1100 ppm F as sodium fluoride (positive control) , 0 ppm F (placebo, negative control)
  Interventions: Drug: 0 ppm F (placebo, negative control); Drug: 1100 ppm F as sodium fluoride (positive control); Drug: 1100 ppm F as sodium fluoride Test Product
- Test-Placebo-Positive (Other): Crossover design - Cleaning, 2-3 day non-F dentifrice, Period 1 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 2 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 3 product for 2 weeks. Product sequence: 1100 ppm F as sodium fluoride Test Product, 0 ppm F (placebo, negative control),1100 ppm F as sodium fluoride (positive control)
  Interventions: Drug: 0 ppm F (placebo, negative control); Drug: 1100 ppm F as sodium fluoride (positive control); Drug: 1100 ppm F as sodium fluoride Test Product
- Positive-Test-Placebo (Other): Crossover design - Cleaning, 2-3 day non-F dentifrice, Period 1 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 2 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 3 product for 2 weeks. Product sequence: 1100 ppm F as sodium fluoride (positive control), 1100 ppm F as sodium fluoride Test Product, 0 ppm F (placebo, negative control)
  Interventions: Drug: 0 ppm F (placebo, negative control); Drug: 1100 ppm F as sodium fluoride (positive control); Drug: 1100 ppm F as sodium fluoride Test Product
- Positive-Placebo-Test (Other): Crossover design - Cleaning, 2-3 day non-F dentifrice, Period 1 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 2 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 3 product for 2 weeks. Product sequence: 1100 ppm F as sodium fluoride (positive control), 0 ppm F (placebo, negative control), 1100 ppm F as sodium fluoride Test Product
  Interventions: Drug: 0 ppm F (placebo, negative control); Drug: 1100 ppm F as sodium fluoride (positive control); Drug: 1100 ppm F as sodium fluoride Test Product
- Placebo-Test-Positive (Other): Crossover design - Cleaning, 2-3 day non-F dentifrice, Period 1 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 2 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 3 product for 2 weeks. Product sequence: 0 ppm F (placebo, negative control), 1100 ppm F as sodium fluoride Test Product,1100 ppm F as sodium fluoride (positive control)
  Interventions: Drug: 0 ppm F (placebo, negative control); Drug: 1100 ppm F as sodium fluoride (positive control); Drug: 1100 ppm F as sodium fluoride Test Product
- Placebo-Positive-Test (Other): Crossover design - Cleaning, 2-3 day non-F dentifrice, Period 1 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 2 product for 2 weeks, 4-5 day washout, cleaning, 2-3 day non-F dentifrice, Period 3 product for 2 weeks. Product sequence: 0 ppm F (placebo, negative control),1100 ppm F as sodium fluoride (positive control), 1100 ppm F as sodium fluoride Test Product
  Interventions: Drug: 0 ppm F (placebo, negative control); Drug: 1100 ppm F as sodium fluoride (positive control); Drug: 1100 ppm F as sodium fluoride Test Product

INTERVENTIONS:
Drug: 0 ppm F (placebo, negative control) — • Each subject will use this product during one of the three treatment periods in the crossover study design.
  Other Names: Tom's of Maine Silly Strawberry
Drug: 1100 ppm F as sodium fluoride (positive control) — • Each subject will use this product during one of the three treatment periods in the crossover study design.
  Other Names: Crest Cavity Protection Toothpaste
Drug: 1100 ppm F as sodium fluoride Test Product — • Each subject will use this product during one of the three treatment periods in the crossover study design.
  Other Names: Pronamel Daily Protection

SUMMARY:
The purpose of this study is to compare the remineralization potential of an optimized fluoride dentifrice to a control fluoride dentifrice in an in situ caries model.

DETAILED DESCRIPTION:
This will be a double blind, single center, 3-way crossover design study. Two to three days before the start of each treatment period the subjects will have their teeth cleaned to remove all accessible plaque and calculus and will be provided with a non-fluoride dentifrice to use until their next visit. At the beginning of each testing period, two gauze-covered 4 mm round partially demineralized bovine enamel specimens will be placed in the buccal surface of two posterior denture teeth (the specimen site may extend into the buccal flange area, if needed) of the same side of the partial denture. Once specimens are placed, subjects will wear their partial dentures twenty-four hours a day and use their assigned toothpaste twice daily, as instructed, until their next visit. Specimens will be removed after two weeks, and the subjects will undergo at least a four- to five-day washout period followed by another cleaning and two to three day lead in period. This process will be repeated until all subjects have used all three test products. Changes in the mineral content of the enamel specimens will be assessed using surface microhardness (SMH) and transverse microradiography (TMR). Enamel fluoride uptake (EFU) will be determined using the microdrill enamel biopsy technique. In addition, the net acid resistance (NAR) and the comparative acid resistance (CAR) of the demineralized enamel specimens will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. provide voluntary, written informed consent;
2. be between 18 and 85 years old;
3. understand and be willing, able and likely to comply with all study procedures and restrictions;
4. be wearing a removable mandibular partial denture with sufficient room to accommodate two 4 mm round specimens in the buccal surface of two posterior denture teeth on the same side;
5. be willing and capable of wearing their removable partial denture 24 hours a day for three (3), two-week treatment periods;
6. be willing to allow study personnel to drill specimen sites in two denture teeth in the posterior section of one side of their lower partial denture, which may extend into the buccal flange area below the teeth;
7. be in good medical and dental health with no active caries or periodontal disease; NOTE: subjects presenting at screening with caries may continue in the study if their carious lesions are restored prior to beginning treatment 1; and
8. have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate ≥ 0.2 mL/min; gum base stimulated whole saliva flow rate ≥ 0.8 mL/min).

Exclusion Criteria:

1. currently be pregnant, intending to become pregnant during the study period or breast feeding;
2. currently have any medical condition that could be expected to interfere with the subject's safety during the study period;
3. currently be taking antibiotics or have taken antibiotics in the two weeks prior to the beginning treatment 1;
4. known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients;
5. have participated in another clinical study or receipt of an investigational drug within 30 days of beginning treatment 1; or
6. be taking fluoride supplements, required to use a fluoride mouthrinse or have received a professional fluoride treatment in the two weeks preceding specimen placement.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domenick Zero, DDS, MS, Principal Investigator — Indiana University; Anderson Hara, DDS, PhD, Principal Investigator — Indiana University; Frank Lippert, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of dentistry, Oral Health Research institute 415 Lansing Street, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clinical Aspects of De/Remineralization of Teeth. Proceedings of Models Conference 1994. Rochester, New York, June 11-14, 1994. Adv Dent Res. 1995 Nov;9(3):169-340. No abstract available. PMID 8615941
- [Background] Corpron RE, Clark JW, Tsai A, More FG, Merrill DF, Kowalski CJ, Tice TR, Rowe CE. Intraoral effects of a fluoride-releasing device on acid-softened enamel. J Am Dent Assoc. 1986 Sep;113(3):383-8. doi: 10.14219/jada.archive.1986.0202. PMID 3463611
- [Background] Featherstone JD, Mellberg JR. Relative rates of progress of artificial carious lesions in bovine, ovine and human enamel. Caries Res. 1981;15(1):109-14. doi: 10.1159/000260508. No abstract available. PMID 6937246
- [Background] Cate JM, Arends J. Remineralization of artificial enamel lesions in vitro. Caries Res. 1977;11(5):277-86. doi: 10.1159/000260279. No abstract available. PMID 18285
- [Background] Koulourides T, Phantumvanit P, Munksgaard EC, Housch T. An intraoral model used for studies of fluoride incorporation in enamel. J Oral Pathol. 1974;3(4):185-96. doi: 10.1111/j.1600-0714.1974.tb01710.x. No abstract available. PMID 4219029
- [Background] Lippert F, Butler A, Lynch RJ. Characteristics of methylcellulose acid gel lesions created in human and bovine enamel. Caries Res. 2013;47(1):50-5. doi: 10.1159/000343164. Epub 2012 Oct 25. PMID 23108261
- [Background] Lippert F, Hara AT. Fluoride dose-response of human and bovine enamel caries lesions under remineralizing conditions. Am J Dent. 2012 Aug;25(4):205-9. PMID 23082383
- [Background] Lippert F, Lynch RJ. Comparison of Knoop and Vickers surface microhardness and transverse microradiography for the study of early caries lesion formation in human and bovine enamel. Arch Oral Biol. 2014 Jul;59(7):704-10. doi: 10.1016/j.archoralbio.2014.04.005. Epub 2014 Apr 21. PMID 24798979
- [Background] Marinho VC, Higgins JP, Sheiham A, Logan S. Fluoride toothpastes for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2003;2003(1):CD002278. doi: 10.1002/14651858.CD002278. PMID 12535435
- [Background] Mellberg JR. Hard-tissue substrates for evaluation of cariogenic and anti-cariogenic activity in situ. J Dent Res. 1992 Apr;71 Spec No:913-9. doi: 10.1177/002203459207100S25. PMID 1592986
- [Background] Proskin HM, Chilton NW, Kingman A. Interim report of the ad hoc committee for the consideration of statistical concerns related to the use of intra-oral models in submissions for product claims approval to the American Dental Association. J Dent Res. 1992 Apr;71 Spec No:949-52. doi: 10.1177/002203459207100S31. PMID 1592992
- [Background] Sakkab NY, Cilley WA, Haberman JP. Fluoride in deciduous teeth from an anti-caries clinical study. J Dent Res. 1984 Oct;63(10):1201-5. doi: 10.1177/00220345840630100601. PMID 6592201
- [Background] Twetman S, Axelsson S, Dahlgren H, Holm AK, Kallestal C, Lagerlof F, Lingstrom P, Mejare I, Nordenram G, Norlund A, Petersson LG, Soder B. Caries-preventive effect of fluoride toothpaste: a systematic review. Acta Odontol Scand. 2003 Dec;61(6):347-55. doi: 10.1080/00016350310007590. PMID 14960006
- [Background] Walsh T, Worthington HV, Glenny AM, Appelbe P, Marinho VC, Shi X. Fluoride toothpastes of different concentrations for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD007868. doi: 10.1002/14651858.CD007868.pub2. PMID 20091655
- [Background] White DJ. Use of synthetic polymer gels for artificial carious lesion preparation. Caries Res. 1987;21(3):228-42. doi: 10.1159/000261026. No abstract available. PMID 3471346
- [Background] Zero DT. In situ caries models. Adv Dent Res. 1995 Nov;9(3):214-30; discussion 231-4. doi: 10.1177/08959374950090030501. PMID 8615944
- [Background] Zero DT, Rahbek I, Fu J, Proskin HM, Featherstone JD. Comparison of the iodide permeability test, the surface microhardness test, and mineral dissolution of bovine enamel following acid challenge. Caries Res. 1990;24(3):181-8. doi: 10.1159/000261263. PMID 2364403

RESULTS

PARTICIPANT FLOW:
Period: Crossover Period 1
Arm/Group | Test-Positive-Placebo | Test-Placebo-Positive | Positive-Test-Placebo | Positive-Placebo-Test | Placebo-Test-Positive | Placebo-Positive-Test
Started | 9 | 8 | 9 | 9 | 8 | 9
Completed | 9 | 8 | 8 | 9 | 7 | 9
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 1 | 0
Period: Washout Between Periods 1 and 2
Arm/Group | Test-Positive-Placebo | Test-Placebo-Positive | Positive-Test-Placebo | Positive-Placebo-Test | Placebo-Test-Positive | Placebo-Positive-Test
Started | 9 | 8 | 8 | 9 | 7 | 9
Completed | 9 | 7 | 8 | 9 | 7 | 9
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Crossover Period 2
Arm/Group | Test-Positive-Placebo | Test-Placebo-Positive | Positive-Test-Placebo | Positive-Placebo-Test | Placebo-Test-Positive | Placebo-Positive-Test
Started | 9 | 7 | 8 | 9 | 7 | 9
Completed | 9 | 6 | 7 | 9 | 7 | 9
Not Completed | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — broken denture | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout Between Periods 2 and 3
Arm/Group | Test-Positive-Placebo | Test-Placebo-Positive | Positive-Test-Placebo | Positive-Placebo-Test | Placebo-Test-Positive | Placebo-Positive-Test
Started | 9 | 6 | 7 | 9 | 7 | 9
Completed | 9 | 6 | 7 | 9 | 7 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover Period 3
Arm/Group | Test-Positive-Placebo | Test-Placebo-Positive | Positive-Test-Placebo | Positive-Placebo-Test | Placebo-Test-Positive | Placebo-Positive-Test
Started | 9 | 6 | 7 | 9 | 7 | 9
Completed | 9 | 6 | 7 | 9 | 7 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This was a three-way crossover design:
  0 ppm F (placebo, negative control;1100 ppm F as sodium fluoride (positive control); 1100 ppm F as sodium fluoride Test Product
Arm/Group | All Study Participants
Number analyzed (Participants) | 52
Age, Continuous [Mean (Full Range); unit: years] | 70 [49 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 32
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Percent Surface Microhardness Recovery (%SMH Recovery)
Description: The SMH test was used to assess changes in the mineral status of partially demineralized enamel specimens.
  %SMH Recovery = (D1-R)/(D1-B) ×100 B = indentation length (µm) of sound enamel specimen at baseline D1 = indentation length (µm) after in vitro demineralization R = indentation length (µm) after intra-oral exposure.
Time Frame: at the end of each two-week treatment per
Population: Analyses were performed using all available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Surface Microhardness Recovery
Groups:
- 0 Ppm F (Placebo); 1100 Ppm F as Sodium Fluoride (Positive Control); 1100 Ppm F as Sodium Fluoride Test Product: Each subject used this product during one of the three treatment periods in the crossover study design.
Arm/Group | 0 Ppm F (Placebo) | 1100 Ppm F as Sodium Fluoride (Positive Control) | 1100 Ppm F as Sodium Fluoride Test Product
Number analyzed (Participants) | 47 | 48 | 49
Percent Surface Microhardness Recovery | 24.4 [19.3 to 29.5] | 51.6 [46.5 to 56.7] | 51.5 [46.5 to 56.6]
Statistical Analysis 1: Comparison: 1100 Ppm F as Sodium Fluoride (Positive Control) vs 1100 Ppm F as Sodium Fluoride Test Product; Based on previous studies we estimate the standard deviation of the differences between treatments in the crossover model to be 20 for % SMH recovery. With a sample size of 58 subjects completing the study, the study had 80% power to detect a difference between any two treatments of 7.5 for % SMH recovery, assuming two-sided tests each conducted at a 5% significance level; Test type: Superiority; p = 0.986, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; Analysis of variance models (ANOVA) suitable for a crossover study, with random effect for subject and fixed effects for study period and product; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-5.5 to 5.4] — Difference calculated as Test-Positive Control
Statistical Analysis 2: Comparison: 0 Ppm F (Placebo) vs 1100 Ppm F as Sodium Fluoride Test Product; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 27.2, 95% CI 2-sided [21.7 to 32.6] — Difference calculated as Test-Placebo
Statistical Analysis 3: Comparison: 0 Ppm F (Placebo) vs 1100 Ppm F as Sodium Fluoride (Positive Control); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 27.2, 95% CI 2-sided [21.7 to 32.7] — Difference calculated as Positive Control-Placebo

2. Secondary Outcome: Enamel Fluoride Uptake (µg F/cm2)
Description: The microdrill enamel biopsy technique will be used to analyze the fluoride content of the partially demineralized enamel specimens. Each enamel specimen will be mounted perpendicular to the long axis of a drill bit attached to a specially designed microdrill and drilled to a depth of ~100 µm through the entire lesion (four cores per specimen). The diameter of the drill hole will be determined using a calibrated microscope interfaced with an image analysis system. The amount of fluoride-uptake by enamel will be calculated based on the amount of fluoride divided by the area of the enamel cores and expressed as µg F/cm2
Time Frame: at the end of each two-week treatment period
Population: Analyses were performed using all available data.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µg F/cm2
Groups:
- 0 Ppm F (Placebo, Negative Control); 1100 Ppm F as Sodium Fluoride (Positive Control); 1100 Ppm F as Sodium Fluoride Test Product: Each subject used this product during one of the three treatment periods in the crossover study design.
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 1100 Ppm F as Sodium Fluoride (Positive Control) | 1100 Ppm F as Sodium Fluoride Test Product
Number analyzed (Participants) | 47 | 48 | 49
µg F/cm2 | 1.99 [1.72 to 2.30] | 10.32 [8.93 to 11.93] | 11.45 [9.92 to 13.22]
Statistical Analysis 1: Comparison: 1100 Ppm F as Sodium Fluoride (Positive Control) vs 1100 Ppm F as Sodium Fluoride Test Product; analyzed as log(EFU); Test type: Superiority; p = 0.230, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 1.11, 95% CI 2-sided [0.93 to 1.32] — Ratio calculated as Test/Positive Control
Statistical Analysis 2: Comparison: 0 Ppm F (Placebo, Negative Control) vs 1100 Ppm F as Sodium Fluoride Test Product; analyzed as log(EFU); Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 5.77, 95% CI 2-sided [4.86 to 6.85] — Ratio calculated as Test/Placebo
Statistical Analysis 3: Comparison: 0 Ppm F (Placebo, Negative Control) vs 1100 Ppm F as Sodium Fluoride (Positive Control); analyzed as log(EFU); Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 5.20, 95% CI 2-sided [4.37 to 6.18] — Ratio calculated as Positive Control/Placebo

3. Secondary Outcome: Percent Net Acid Resistance
Description: % Net Acid Resistance = [(D1-D2) / (D1-B)] * 100 B= Indentation length (µm) of sound enamel at baseline D1= Indentation length (µm) after first in vitro demineralization D2= Indentation length (µm) after second in vitro demineralization
Time Frame: at the end of each two-week treatment period
Population: Analyses were performed using all available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Net Acid Resistance
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 1100 Ppm F as Sodium Fluoride (Positive Control) | 1100 Ppm F as Sodium Fluoride Test Product
Number analyzed (Participants) | 47 | 48 | 49
Percent Net Acid Resistance | 2.6 [-2.3 to 7.4] | 34.3 [29.5 to 39.1] | 37.4 [32.6 to 42.1]
Statistical Analysis 1: Comparison: 1100 Ppm F as Sodium Fluoride (Positive Control) vs 1100 Ppm F as Sodium Fluoride Test Product; Test type: Superiority; p = 0.272, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-2.5 to 8.6] — Difference calculated as Test-Positive Control
Statistical Analysis 2: Comparison: 0 Ppm F (Placebo, Negative Control) vs 1100 Ppm F as Sodium Fluoride Test Product; Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 34.8, 95% CI 2-sided [29.3 to 40.3] — Difference calculated as Test-Placebo
Statistical Analysis 3: Comparison: 0 Ppm F (Placebo, Negative Control) vs 1100 Ppm F as Sodium Fluoride (Positive Control); Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 31.7, 95% CI 2-sided [26.2 to 37.3] — Difference calculated as Positive Control-Placebo

4. Secondary Outcome: Percentage Comparative Acid Resistance
Description: % Comparative Acid Resistance = [(D2-R) / (D1-B)] * 100 B= Indentation length (µm) of sound enamel at baseline R= Indentation length (µm) of enamel after in situ remineralization D1= Indentation length (µm) after first in vitro demineralization D2= Indentation length (µm) after second in vitro demineralization
Time Frame: at the end of each two-week treatment period
Population: Analyses were performed using all available data.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percentage Comparative Acid Resistance
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 1100 Ppm F as Sodium Fluoride (Positive Control) | 1100 Ppm F as Sodium Fluoride Test Product
Number analyzed (Participants) | 47 | 48 | 49
Percentage Comparative Acid Resistance | 20.27 [16.26 to 24.43] | 16.40 [12.55 to 20.39] | 13.51 [9.78 to 17.36]
Statistical Analysis 1: Comparison: 1100 Ppm F as Sodium Fluoride (Positive Control) vs 1100 Ppm F as Sodium Fluoride Test Product; analyzed as log(%CAR+100); Test type: Superiority; p = 0.191, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 1.11, 95% CI 2-sided [0.93 to 1.32] — Ratio calculated as Test/Positive Control
Statistical Analysis 2: Comparison: 0 Ppm F (Placebo, Negative Control) vs 1100 Ppm F as Sodium Fluoride Test Product; analyzed as log(%CAR+100); Test type: Superiority; p = 0.003, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 0.94, 95% CI 2-sided [0.91 to 0.98] — Ratio calculated as Test/Placebo
Statistical Analysis 3: Comparison: 0 Ppm F (Placebo, Negative Control) vs 1100 Ppm F as Sodium Fluoride (Positive Control); analyzed as log(%CAR+100); Test type: Superiority; p = 0.092, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 0.97, 95% CI 2-sided [0.93 to 1.01] — Ratio calculated as Positive Control/Placebo

5. Secondary Outcome: Integrated Mineral Loss (∆Z)
Description: ∆Z= [(lesion depth x 87) - area under the curve*] calculated using Transverse Microradiography software program
Time Frame: at the end of each two-week treatment period
Population: Analyses were performed using all available data.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Integrated Mineral Loss (∆Z)
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 1100 Ppm F as Sodium Fluoride (Positive Control) | 1100 Ppm F as Sodium Fluoride Test Product
Number analyzed (Participants) | 47 | 48 | 49
Integrated Mineral Loss (∆Z) | 998 [917 to 1087] | 703 [646 to 765] | 708 [651 to 770]
Statistical Analysis 1: Comparison: 1100 Ppm F as Sodium Fluoride (Positive Control) vs 1100 Ppm F as Sodium Fluoride Test Product; analyzed as log(∆Z); Test type: Superiority; p = 0.905, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 1.01, 95% CI 2-sided [0.90 to 1.13] — Ratio calculated as Test/Positive Control
Statistical Analysis 2: Comparison: 0 Ppm F (Placebo, Negative Control) vs 1100 Ppm F as Sodium Fluoride Test Product; analyzed as log(∆Z); Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 0.71, 95% CI 2-sided [0.63 to 0.80] — Ratio calculated as Test/Placebo
Statistical Analysis 3: Comparison: 0 Ppm F (Placebo, Negative Control) vs 1100 Ppm F as Sodium Fluoride (Positive Control); analyzed as log(∆Z); Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 0.70, 95% CI 2-sided [0.63 to 0.79] — Ratio calculated as Positive Control/Placebo

6. Secondary Outcome: Lesion Depth (µm)
Description: Lesion Depth - L (83% mineral i.e. 95% of the mineral content of sound enamel) determined using Transverse Microradiography software program
Time Frame: at the end of each two-week treatment period
Population: Analyses were performed using all available data.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µm
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 1100 Ppm F as Sodium Fluoride (Positive Control) | 1100 Ppm F as Sodium Fluoride Test Product
Number analyzed (Participants) | 47 | 48 | 49
µm | 40.5 [37.2 to 44.1] | 31.2 [28.7 to 33.9] | 30.6 [28.1 to 33.2]
Statistical Analysis 1: Comparison: 1100 Ppm F as Sodium Fluoride (Positive Control) vs 1100 Ppm F as Sodium Fluoride Test Product; analyzed as log(lesion depth); Test type: Superiority; p = 0.721, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 0.98, 95% CI 2-sided [0.88 to 1.09] — Ratio calculated as Test/Positive Control
Statistical Analysis 2: Comparison: 0 Ppm F (Placebo, Negative Control) vs 1100 Ppm F as Sodium Fluoride Test Product; analyzed as log(lesion depth); Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 0.75, 95% CI 2-sided [0.68 to 0.84] — Ratio calculated as Test/Placebo
Statistical Analysis 3: Comparison: 0 Ppm F (Placebo, Negative Control) vs 1100 Ppm F as Sodium Fluoride (Positive Control); analyzed as log(lesion depth); Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Ratio of Means = 0.77, 95% CI 2-sided [0.69 to 0.86] — Ratio calculated as Positive Control/Placebo

7. Secondary Outcome: Maximum Mineral Density at the Surface-zone (SZmax)
Description: SZmax was determined using Transverse Microradiography software program
Time Frame: at the end of each two-week treatment period
Population: Analyses were performed using all available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Maximum mineral density at the surface-z
Arm/Group | 0 Ppm F (Placebo) | 1100 Ppm F as Sodium Fluoride (Positive Control) | 1100 Ppm F as Sodium Fluoride Test Product
Number analyzed (Participants) | 47 | 48 | 49
Maximum mineral density at the surface-z | 59.26 [57.40 to 61.12] | 66.17 [64.32 to 68.01] | 65.61 [63.79 to 67.44]
Statistical Analysis 1: Comparison: 1100 Ppm F as Sodium Fluoride (Positive Control) vs 1100 Ppm F as Sodium Fluoride Test Product; Test type: Superiority; p = 0.647, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-2.95 to 1.84] — Difference calculated as Test-Positive Control
Statistical Analysis 2: Comparison: 0 Ppm F (Placebo) vs 1100 Ppm F as Sodium Fluoride Test Product; Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.35, 95% CI 2-sided [3.95 to 8.75] — Difference calculated as Test-Placebo
Statistical Analysis 3: Comparison: 0 Ppm F (Placebo) vs 1100 Ppm F as Sodium Fluoride (Positive Control); Test type: Superiority; p < 0.001, Mixed Models Analysis — No alpha-level adjustments for multiple comparisons adjustments were applied; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.90, 95% CI 2-sided [4.49 to 9.31] — Difference calculated as Positive Control-Placebo

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | 0 Ppm F (Placebo) | 1100 Ppm F as Sodium Fluoride (Positive Control) | 1100 Ppm F as Sodium Fluoride Test Product
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/52 | 1/52
Other Adverse Events (participants affected / at risk) | 23/52 | 16/52 | 19/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0 Ppm F (Placebo) (N=52) | 1100 Ppm F as Sodium Fluoride (Positive Control) (N=52) | 1100 Ppm F as Sodium Fluoride Test Product (N=52)
Bowel Obstructiion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Bowel obstruction due to adhesions. The subject had abdominal distress with nausea and vomiting which required hospital admission and surgery from which the subject fully recovered.
Migraine vestibulaire (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Subject had a history of migraines and experienced severe migraine that required hospitalization. The subject received treatment with Meclizine and all symptoms resolved in a few days.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0 Ppm F (Placebo) (N=52) | 1100 Ppm F as Sodium Fluoride (Positive Control) (N=52) | 1100 Ppm F as Sodium Fluoride Test Product (N=52)
Flu (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cold Sweats (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lack of balance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Common cold (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 2 (2)
Erythema Mandibular Ridge (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) — Erythema due to partial denture friction
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Prolonged Post Operative Lleus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry, cracked lower lip (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Burning Sensation Oral Cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Transient Sour Sensation in Oral Cavity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Transient Sour Sensation in Mandibular Posterior Area, while eating. bilateral
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica Nerve Pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Sciatica, left side pain
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fractured Metal Frame of the Mandibular Partial (Product Issues) | 0 (0) | 0 (0) | 1 (1) — The metal framework of the subjects partial denture appliance broke.
Earache (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Oral ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) — Oral ulcer due to partial denture friction
Herpetic Lesion Upper Lip (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dry and Chapped Lower Lip (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Swollen Lower Lip (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tenderness Oral Cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Tenderness Mandibular Left Side Edentulous pre-molar area from Partial Denture Friction
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Basel cell carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Basel cell carcinoma on the skin of left thigh treated with surgical excision
Bladder Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Worsening of the lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema, Hard palate (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Erythema, Hard palate 3X8mm due to food burn
Pain anterior gingiva (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Pain from wearing partial at night with C-PAP mask on anterior gingiva
Erythema buccal mucosa due to cheek bite (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) — Erythema on left side of buccal mucosa posterior 3mmX3mm due to cheek bite
Body ache from shingle vaccine (General disorders) | 1 (1) | 0 (0) | 0 (0)
Worsening of COPD symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Worsening of Asthma symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Muscle Strain - Left shoulder blade
Worsening of Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT06010732/Prot_SAP_000.pdf